CLINICAL TRIAL: NCT06532942
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Nintedanib Inhalation Powder (MNKD-201) in Healthy Volunteers
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of MKND-201 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKC-NI-001
Record Dates: First submitted 2024-07-26; First posted 2024-08-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This first-in-human trial will be conducted in healthy adult volunteers and will investigate the safety, tolerability, and PK of MNKD-201. MNKD-201 will be evaluated over a range of doses, first in a SAD phase (Part A) and then in a MAD phase (Part B), to inform doses for further evaluation in a subsequent trial. Approximately 40 participants will be enrolled into 1 of 3 SAD cohorts and 2 MAD cohorts, 8 participants per cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- (Part A) MKND-201 SAD (Experimental): Part A involves a Single Ascending Dose (SAD) study with three cohorts. In each cohort, participants will receive a single dose of MKND-201 or placebo for one day. The doses will be categorized as Target Dose, High Dose, and Very High Dose. Allocation is randomized and double-blind, maintaining a ratio of 3:1 (MKND-201:placebo). Participants will use a breath-powered inhaler, which aerosolizes the powder for lung delivery
  Interventions: Drug: (Part A) MKND-201
- (Part B) MKND-201 MAD (Experimental): Part B involves a Multiple Ascending Dose (MAD) study with two cohorts. In each cohort, participants will receive MKND-201 or placebo twice daily (BID) at either the Target Dose or High Dose. Allocation is randomized 3:1 (MKND-201:placebo) and double-blind. Participants will use a breath-powered inhaler, which aerosolizes the powder for lung delivery
  Interventions: Drug: (Part B) MKND-201
- Placebo (Placebo Comparator): Administered as a single dose or BID using the same number of cartridges as MKND-201 participants in the same cohort
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: (Part A) MKND-201 — Participants will receive single ascending doses (Target Dose, High Dose, and Very High Dose) of MKND-201 or placebo administered via oral inhalation on Day 1
  Arms: (Part A) MKND-201 SAD
Drug: Placebo — Participants will receive matching placebo across Part A and Part B of the study.
  Arms: Placebo
Drug: (Part B) MKND-201 — Participants will receive multiple ascending doses (Target Dose and High Dose) of MKND-201 or placebo administered via oral inhalation, twice daily, from Day 1 to Day 7
  Arms: (Part B) MKND-201 MAD

SUMMARY:
MKC-NI-001 is a Phase 1, first-in-human, randomized, double-blind, placebo-controlled study of nintedanib inhalation powder (MNKD-201) in healthy adult volunteers. The trial consists of a Single Ascending Dose (SAD), followed by a Multiple Ascending Dose (MAD) with a primary objective to evaluate the safety, tolerability, and pharmacokinetics (PK) of MNKD-201 compared to placebo in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Is ≥40 and ≤65 years of age at the time of signing the informed consent form.
* Has a negative urine test for selected drugs of abuse and negative alcohol test at screening and upon admission to the CRU on Day -1. Note: Participants should not consume poppy seeds within 24 hours before urine drug screening because this can falsify the results of the opiate urine drug test.
* Is willing to adhere to the restrictions and requirements specified in the protocol.
* Has a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test (i.e., the virus that causes COVID-19) on Day -1.
* Is capable of performing spirometry, as required by the study procedures.

Key Exclusion Criteria:

* Has a history of significant lung disease (e.g., pulmonary fibrosis, cystic fibrosis, COPD, emphysema, chronic pulmonary infection, recent upper or lower respiratory tract infection in the prior 8 weeks, history of lung surgery or procedure, etc.)
* Has endocrine, thyroid, or respiratory disease, diabetes mellitus, coronary heart disease, GI disease, or history of any psychotic mental illness.
* Has a history of hepatic disease or has abnormal liver function tests (i.e., aspartate aminotransferase [AST] > 1.5 × upper limit of normal [ULN] or alanine aminotransferase [ALT] > 1.5 × ULN) at screening.
* Has renal impairment (estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73 m2), as calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), at screening.
* Has any history of pulmonary malignancy.
* Has a history of substance abuse or dependency or history of recreational drug use over the last 2 years (by self-declaration).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
(Part A) Incidence of inhaled intolerability | Up to Day 9 (+/- 3 days)
  Incidence of inhaled intolerability (prevalence of cough, dyspnea, bronchospasm, and dysgeusia)
(Part B) Incidence of inhaled intolerability | Up to Day 15 (+/- 3 days)
  Incidence of inhaled intolerability (prevalence of cough, dyspnea, bronchospasm, and dysgeusia)
(Part A) Incidence of participants with reductions in FEV1 ≥ 15% from baseline at any time postdose | Up to Day 9 (+/- 3 days)
  Incidence of participants with reductions in FEV1 ≥ 15% from baseline at any time postdose
(Part B) Incidence of participants with reductions in FEV1 ≥ 15% from baseline at any time postdose | Up to Day 15 (+/- 3 days)
  Incidence of participants with reductions in FEV1 ≥ 15% from baseline at any time postdose
(Part A) Incidence of participants with reductions in FEV1 ≥ 15% following administration of a dose of study drug, compared to the corresponding predose measurement | Up to Day 9 (+/- 3 days)
  Incidence of participants with reductions in FEV1 ≥ 15% following administration of a dose of study drug, compared to the corresponding predose measurement
(Part B) Incidence of participants with reductions in FEV1 ≥ 15% following administration of a dose of study drug, compared to the corresponding predose measurement | Up to Day 15 (+/- 3 days)
  Incidence of participants with reductions in FEV1 ≥ 15% following administration of a dose of study drug, compared to the corresponding predose measurement
(Part A) Incidence of treatment-emergent adverse events (TEAEs) | Up to Day 9 (+/- 3 days)
  Incidence, severity, duration, relationship to study drug, and outcome of treatment-emergent adverse events (TEAEs)
(Part B) Incidence of treatment-emergent adverse events (TEAEs) | Up to Day 15 (+/- 3 days)
  Incidence, severity, duration, relationship to study drug, and outcome of treatment-emergent adverse events (TEAEs)
(Part A) Incidence of serious adverse events (SAEs) | Up to Day 9 (+/- 3 days)
  Incidence, severity, duration, relationship to study drug, and outcome of serious adverse events (SAEs)
(Part B) Incidence of serious adverse events (SAEs) | Up to Day 15 (+/- 3 days)
  Incidence, severity, duration, relationship to study drug, and outcome of serious adverse events (SAEs)
(Part A) Incidence of abnormal clinically significant vital signs | Up to Day 9 (+/- 3 days)
  Incidence of abnormal clinically significant vital signs (heart rate, blood pressure, respiratory rate, oxygen saturation rate, and body temperature)
(Part B) Incidence of abnormal clinically significant vital signs | Up to Day 15 (+/- 3 days)
  Incidence of abnormal clinically significant vital signs (heart rate, blood pressure, respiratory rate, oxygen saturation rate, and body temperature)
(Part A) Changes from baseline in liver enzymes and bilirubin | Up to Day 9 (+/- 3 days)
  Changes from baseline in liver enzymes and bilirubin
(Part B) Changes from baseline in liver enzymes and bilirubin | Up to Day 15 (+/- 3 days)
  Changes from baseline in liver enzymes and bilirubin
(Part A) Changes from baseline in coagulation parameters, INR and aPTT | Up to Day 9 (+/- 3 days)
  Changes from baseline in coagulation parameters - international normalized ratio (INR) and activated partial thromboplastin time (aPTT)
(Part B) Changes from baseline in coagulation parameters, INR and aPTT | Up to Day 15 (+/- 3 days)
  Changes from baseline in coagulation parameters - international normalized ratio (INR) and activated partial thromboplastin time (aPTT)

SECONDARY OUTCOMES:
(Part A) Maximum plasma MNKD-201 concentration (Cmax) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Maximum plasma MNKD-201 concentration (Cmax)
(Part B) Maximum plasma MNKD-201 concentration (Cmax) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) Maximum plasma MNKD-201 concentration (Cmax)
(Part A) Time to maximum concentration (Tmax) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Time to maximum concentration (Tmax)
(Part B) Time to maximum concentration (Tmax) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) Time to maximum concentration (Tmax)
(Part A) Terminal elimination half-life (t½) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Terminal elimination half-life (t½)
(Part B) Terminal elimination half-life (t½) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) Terminal elimination half-life (t½)
(Part A) Area under the plasma concentration-time curve (AUC) from time zero (from the start of inhalation time) to the last measurable concentration (AUC0-t) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Area under the plasma concentration-time curve (AUC) from time zero (from the start of inhalation time) to the last measurable concentration (AUC0-t)
(Part A) Area under the plasma concentration-time curve (AUC) from time zero (from the start of inhalation time) to the last measurable concentration (AUC0-t) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part A) Area under the plasma concentration-time curve (AUC) from time zero (from the start of inhalation time) to the last measurable concentration (AUC0-t)
(Part A) AUC from time zero (time of first inhalation) to infinity (AUC0-∞) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) AUC from time zero (time of first inhalation) to infinity (AUC0-∞)
(Part B) AUC from time zero (time of first inhalation) to infinity (AUC0-∞) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) AUC from time zero (time of first inhalation) to infinity (AUC0-∞)
(Part A) Apparent terminal elimination rate constant (Kel) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Apparent terminal elimination rate constant (Kel)
(Part B) Apparent terminal elimination rate constant (Kel) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) Apparent terminal elimination rate constant (Kel)
(Part A) Apparent total body clearance (CL/F) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Apparent total body clearance (CL/F)
(Part B) Apparent total body clearance (CL/F) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) Apparent total body clearance (CL/F)
(Part A) Apparent volume of distribution during the terminal phase (Vz/F) | Day 1, predose and at multiple time points postdose up to Day 2, 24 hours postdose
  (Part A) Apparent volume of distribution during the terminal phase (Vz/F)
(Part B) Apparent volume of distribution during the terminal phase (Vz/F) | Day 1, predose and at multiple time points postdose up to Day 8, 12 hours after last dose on Day 7
  (Part B) Apparent volume of distribution during the terminal phase (Vz/F)
(Part A) Changes in forced expiratory volume in 1 second (FEV1) before and after dosing | predose and 5, 15, 30, 60, 90, and 120 minutes postdose
  (Part A) Changes in forced expiratory volume in 1 second (FEV1) before and after dosing (predose and 5, 15, 30, 60, 90, and 120 minutes postdose)
(Part B) Changes in forced expiratory volume in 1 second (FEV1) before and after dosing | predose and 5, 15, 30, 60, 90, and 120 minutes postdose
  (Part B) Changes in forced expiratory volume in 1 second (FEV1) before and after dosing (predose and 5, 15, 30, 60, 90, and 120 minutes postdose)

CONTACTS AND LOCATIONS:
Locations (1):
- Flourish Research, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No